CLINICAL TRIAL: NCT00773045
Title: Pain Measurement and Pain Management in the ICU
Brief Title: Pain Measurement and Pain Management in the Intensive Care Unit(ICU)
Acronym: PIJNICU2
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: P Bruins, MD, PhD, Department of Anaesthesiology, Intensive Care and Pain Management, St Antonius Hospital
Other Study IDs: PIJNICU2/Z06.11
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Critically Ill Patients
Keywords: pain scores; critically ill patients; ICU; pain management; pain measurement
MeSH Terms: conditions — Agnosia | interventions — Pain Management

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pain training program: ICU Patients treated with or without pain management protocol
  Interventions: Other: A Pain training program and pain measurement

INTERVENTIONS:
Other: A Pain training program and pain measurement — Comparing patients treated with and without analgesia and sedation protocol
  Other Names: pain measurement; pain management

SUMMARY:
The purpose of this study is to evaluate the effect of a pain training program and systematic measurement of pain scores on actual pain levels and the use of analgesics in critically ill patients.

DETAILED DESCRIPTION:
Systematic evaluation of pain, though still not common practice in all ICUs, is recommended in clinical practice guidelines for optimal pain management. Pain is a frequently experienced problem in patients in the Intensive Care Unit(ICU). In search of literature to support the need for introduction of a pain management system and to train the entire health staff in our department little information was found concerning the effects of pain training and pain management systems in the ICU. The small number of available studies may be explained by the difficulty of systematic pain measurement in ICU patients, mainly due to the inability to communicate effectively with these patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ICU of the St. Antonius hospital, >18 years old.

Exclusion Criteria:

* Patients who are suspected to be brain-dead

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients, 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2006-04; Primary Completion 2006-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Pain scores using the numerical rating scale, rated by the attending nurse and by the patient if possible. | 3 times a day

SECONDARY OUTCOMES:
Dose of all pain medication (morphine, paracetamol) per patient | 24 hr
Length of stay in the ICU | ICU stay
Pneumonia | ICU stay
30 day Mortality | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bruins, MD, PhD, Principal Investigator — Department of Anaesthesiology, Intensive Care and Pain Management, St Antonius Hospital, Nieuwegein